CLINICAL TRIAL: NCT02057042
Title: Veteran Peer-Assisted Computerized Cognitive Behavioral Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 13-310
Record Dates: First submitted 2014-01-07; First posted 2014-02-06 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: Depression
Keywords: Peer Support; cCBT; primary care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PS-cCBT (Experimental): peer-assisted computerized CBT
  Interventions: Behavioral: Peer-assisted computerized CBT
- EUC (Active Comparator): Enhanced usual care
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Peer-assisted computerized CBT — Patients in the PS-cCBT intervention will receive usual depression care and will also receive: 1) access to Beating the Blues (BTB), an online cCBT program, 2) support of a peer specialists for 12 weeks, 3) a copy of the Depression Helpbook by Wayne Katon and colleagues
  Arms: PS-cCBT
Behavioral: Enhanced usual care — Patients randomized to EUC will receive the following enhancements: 1) patient education regarding the symptoms of depression and evidence-based depression treatments, 2) a copy of the Depression Helpbook by Wayne Katon and colleagues 3) information about how to access local VA mental health depression treatment resources (groups, individual psychotherapy, etc), and 4) bi-weekly study mailings with depression management tips.
  Arms: EUC

SUMMARY:
The investigators will conduct a randomized clinical trial of Peer-Supported cCBT versus enhanced usual care (EUC) for 330 patients with new episodes of depression in primary care at three VA sites and their associated Community-Based Outpatient Clinics (CBOCs).

DETAILED DESCRIPTION:
Background:

Antidepressant medications and evidence-based psychotherapies are effective treatments for depression. However, antidepressant medication adherence continues to be suboptimal and offering access to and retaining patients in evidence-based psychotherapies for depression is challenging. The VHA has made major efforts to expand access to and capacity for depression focused evidence-based psychotherapies. However in 2012, only 35% of VA patients with depression completed any psychotherapy visit and only 6% completed 8 psychotherapy visits in 14 weeks, a proxy for an adequate trial.

Initiation and engagement in depression treatment may be increased if patients are offered timely access to a highly flexible, evidence-based treatment options, such as a tailored, web-based computerized cognitive-behavioral therapy (cCBT) program. cCBT has sufficient evidence for effectiveness to be a covered benefit in United Kingdom National Health Service, but has much larger effects when it is supported by clinicians or other trusted individuals. VA peer specialists, an increasing workforce in VHA mental health, are ideal candidates to support patients' engagement in depression treatment and in cCBT. Peers have been shown to promote use of Internet self-management tools, and peer specialist support for cCBT may enhance its completion and overall effectiveness through regular "check ins" and also through providing peer specific experiences, such as sharing of lived experiences and modeling of self management and recovery.

Objectives:

We are conducting a Hybrid Type I RCT of Peer-Supported cCBT versus enhanced usual care (EUC) for 330 patients with new episodes of depression in primary care at three VA sites and their associated CBOCs. Our specific aims are to compare PS-cCBT versus enhanced usual care (EUC) on: a) patient symptomatic, functional, and recovery-oriented outcomes, b) depression coping skills, antidepressant medication adherence, and initiation and completion of more intensive traditional psychotherapy (contingent on symptom level). Our secondary aims are to assess patient, peer, and providers' experiences in PS-cCBT versus EUC using mixed methods. Finally, our exploratory aim is to assess potential mediators of improvements in depressive symptoms or functional status.

Methods:

This is a Hybrid I randomized controlled trial (RCT) of peer-supported cCBT compared to enhanced usual care (EUC) among Veterans with new diagnoses of depression in primary care. The cCBT program consists of 8 modules and will be supported by VA peer specialists with weekly contact for 12 weeks. We will assess patient symptomatic, functional and recovery-oriented outcomes at 12 and 24 week following randomization. We will also assess potential mediators of these outcomes. Bivariate and multivariate study analyses will assess the impact of the two study arms at each assessment point and over time.

Status:

Study is currently ongoing, study recruitment and follow-up is active.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for the study if they:

* have new episodes of depression in primary care, defined as those with a new diagnoses of depression and no prior depression diagnoses or antidepressant fills within 120 days of the index date of their depression diagnosis any of three VA study sites or associated CBOCs. Patients must enroll within 90 days of their diagnosis.
* have a current Patient Health Questionnaire (PHQ)-9 score > 10.
* are not receiving mental health care outside of VHA.
* have broadband internet access at home or confirm willingness, ability, and a plan to go to their VA facility to complete cCBT modules.
* have familiarity with email and internet use.
* have stable access to and ability to communicate by telephone.

Exclusion Criteria:

Exclusion criteria for the study will include:

* a diagnosis of schizophrenia, schizoaffective disorder, major depressive disorder (MDD) with psychotic features, or Bipolar I in the past 24 months.
* a positive screen for moderate or severe substance use (AUDIT-C >7).
* an immediate risk of suicide, requiring hospitalization or urgent evaluation (as evidenced by suicidal plan or intent).
* participating in other research studies.
* diagnosis of depression in the past 4 months from a non-VA provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul N Pfeiffer, MD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (3):
- United States (3):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Battle Creek VA Medical Center, Battle Creek, MI, Battle Creek, Michigan
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abraham KM, Nelson CB, Ganoczy D, Zivin K, Brandfon S, Walters H, Cohen JL, Valenstein M. Psychometric analysis of the Mental Health Recovery Measure in a sample of veterans with depression. Psychol Serv. 2016 May;13(2):193-201. doi: 10.1037/ser0000067. PMID 27148954
- [Result] Barry CN, Abraham KM, Weaver KR, Bowersox NW. Innovating team-based outpatient mental health care in the Veterans Health Administration: Staff-perceived benefits and challenges to pilot implementation of the Behavioral Health Interdisciplinary Program (BHIP). Psychol Serv. 2016 May;13(2):148-155. doi: 10.1037/ser0000072. PMID 27148949
- [Derived] Pfeiffer PN, Pope B, Houck M, Benn-Burton W, Zivin K, Ganoczy D, Kim HM, Walters H, Emerson L, Nelson CB, Abraham KM, Valenstein M. Effectiveness of Peer-Supported Computer-Based CBT for Depression Among Veterans in Primary Care. Psychiatr Serv. 2020 Mar 1;71(3):256-262. doi: 10.1176/appi.ps.201900283. Epub 2020 Jan 14. PMID 31931686

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced Usual Care | PS-cCBT
Started | 163 | 167
Completed | 118 | 101
Not Completed | 45 | 66

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | PS-cCBT | Total
Number analyzed (Participants) | 163 | 167 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (15.5) | 51.6 (14.4) | 51.6 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 36 | 65
  Male | 134 | 131 | 265
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 119 | 115 | 234
  Black | 31 | 37 | 68
  Other | 13 | 15 | 28
  Hispanic | 3 | 6 | 9
Education [Count of Participants; unit: Participants]
  High school or less | 37 | 21 | 58
  Some college | 64 | 82 | 146
  College graduate | 61 | 63 | 124

OUTCOME MEASURES:

1. Primary Outcome: Functional Status
Description: Functional status will be measured using the Veterans RAND 12-Item Health Survey (VR-12). Developed from VR-36, VR-12 includes 12 original question items from the VR-36. The questions in this survey correspond to seven different health domains inlcuding general health perceptions, physical functioning, role limitations due to physical and emotional problems, bodily pain, energy/fatigue levels, social functioning and mental health. Answers are summarized into a Physical Component Score (PCS) and a Mental Component Score (MCS) which allows for a comparison between the respondents physical and psychological health status.The VR-12 has somewhat greater precision at the lower end of the health status continuum than the SF-12. The VR-12 has been used in numerous prior VA focused studies. VR-12 MCS component scores are standardized to a mean of 50, with higher scores indicating better mental health and related functioning.
Time Frame: change over time (baseline, 3 months, 6 months)
Population: Numbers analyzed in each time period account for attrition in follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | PS-cCBT
Number analyzed (Participants) | 163 | 167
score on a scale
  Baseline | 32.1 (9.9) | 31.4 (9.7)
  3 months: number analyzed (Participants) | 128 | 108
  3 months | 36.2 (10.3) | 37.3 (11.5)
  6 months: number analyzed (Participants) | 118 | 101
  6 months | 37.1 (11.0) | 40.1 (12.2)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs PS-cCBT; Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Depression Symptoms
Description: Inventory of Depressive Symptoms (IDS) at baseline, 3 months post intervention and 6 months post intervention. The ISD is a 16-item self-report instrument for measuring the severity of depression among individuals. Each item is rated on a four-point scale (0-3), and aggregate scores range from 0 to 27. The IDS has been widely used and shows acceptable reliability, with Cronbach's of 0.86. Severity of depression is scored according to the following ranges: 1-5 (no depression), 6-10 (mild), 11-15 (moderate), 16-20 (severe), and 21-27 (very severe).
Time Frame: change over time (baseline, 3 months, 6 months)
Population: Numbers analyzed in each time period account for attrition in follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | PS-cCBT
Number analyzed (Participants) | 163 | 167
score on a scale
  Baseline | 13.4 (3.6) | 14.0 (3.9)
  3 months: number analyzed (Participants) | 128 | 108
  3 months | 11.7 (4.1) | 11.1 (4.7)
  6 months: number analyzed (Participants) | 118 | 101
  6 months | 11.2 (4.4) | 10.6 (5.1)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs PS-cCBT; Test type: Superiority; p < 0.05, Mixed Models Analysis

3. Primary Outcome: Recovery Orientation
Description: Recovery orientation will be measured using the Recovery Assessment Scale - Short Form (RAS-SF). This 20-item scale is a shorter version of the RAS and has four factors: personal confidence and hope, willingness to ask for help, reliance on others, and no domination by symptoms. The RAS-SF shows evidence for both convergent and discriminate validity when compared to quality of life, social support, and symptomatic scales. The scale is scored by summing all items (or scale items), with 100 being the highest possible overall score. Higher scores indicate greater sense of recovery.
Time Frame: change over time (baseline, 3 months, 6 months)
Population: Numbers analyzed in each time period account for attrition in follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | PS-cCBT
Number analyzed (Participants) | 163 | 167
score on a scale
  Baseline | 69.3 (9.7) | 67.1 (11.1)
  3 months: number analyzed (Participants) | 128 | 108
  3 months | 71.7 (10.5) | 72.6 (13.7)
  6 months: number analyzed (Participants) | 118 | 101
  6 months | 71.1 (11.7) | 74.1 (14.6)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs PS-cCBT; Test type: Superiority; p < 0.05, Mixed Models Analysis

4. Primary Outcome: Quality of Life Enjoyment and Satisfaction
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) is a valid proxy for the longer Quality of Life Enjoyment and Satisfaction (Q-LES) form and will be used to assess quality of life. It consists of 14 items that patients rate on a 5-point scale to indicate their satisfaction with a variety of life domains, including physical health, mood, work, household activities, social relationships, etc. The Q-LES-Q-SF has been shown to have high levels of reliability and has been used in numerous studies of depression, including the National Institute of Mental Health (NIMH) funded STAR*D study. Responses are scored on a 5-point scale, where higher scores indicate better enjoyment and satisfaction with life (possible range 14-70).
Time Frame: change over time (baseline, 3 months, 6 months)
Population: Numbers analyzed in each time period account for attrition in follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | PS-cCBT
Number analyzed (Participants) | 163 | 167
score on a scale
  Baseline | 38.8 (8.7) | 37.7 (8.3)
  3 months: number analyzed (Participants) | 128 | 108
  3 months | 40.5 (9.9) | 41.6 (9.9)
  6 months: number analyzed (Participants) | 118 | 101
  6 months | 41.0 (10.4) | 42.5 (10.7)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs PS-cCBT; Test type: Superiority; p < 0.05, Mixed Models Analysis

5. Secondary Outcome: Cognitive Behavioral Therapy Skills
Description: CBT skills will be assessed using the Cognitive-Behavioral Therapy Skills Questionnaire (CBTSQ). The CBTSQ is a 16-item scale consisting of two factors, Behavioral Activation and Cognitive Restructuring. The scale shows construct validity, appears sensitive to change among patients undergoing CBT treatment, and predicts reduction in depressive symptoms. Scores are summed with a maximum score of 80. Higher scores indicate greater uptake of CBT skills.
Time Frame: change over time (baseline, 3 months, 6 months)
Population: Numbers analyzed in each time period account for attrition in follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | PS-cCBT
Number analyzed (Participants) | 163 | 167
score on a scale
  Baseline | 42.4 (10.2) | 40.4 (11.0)
  3 months: number analyzed (Participants) | 128 | 108
  3 months | 45.1 (10.7) | 46.1 (12.6)
  6 months: number analyzed (Participants) | 118 | 101
  6 months | 45.9 (10.8) | 48.0 (14.3)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs PS-cCBT; Test type: Superiority; p < 0.05, t-test, 2 sided

6. Secondary Outcome: Anxiety
Description: Generalized Anxiety will be measured with the Generalized Anxiety Disorder 7-item (GAD-7). Total score ranges from 0 to 21, with "cut scores" for mild, moderate and severe anxiety. Although originally developed for generalized anxiety disorder symptoms, the GAD-7 has good operating characteristics for detection and severity ratings of panic disorder and social anxiety disorder. Scores are summed with a range of 0-21. Scores represent: 0-5 mild, 6-10 moderate, 11-15 moderate/severe, and 15-21 severe anxiety.
Time Frame: change over time (baseline, 3 months, 6 months)
Population: Numbers analyzed in each time period account for attrition in follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | PS-cCBT
Number analyzed (Participants) | 163 | 167
score on a scale
  Baseline | 11.3 (4.7) | 11.0 (4.3)
  3 months: number analyzed (Participants) | 128 | 108
  3 months | 9.5 (4.8) | 8.8 (5.1)
  6 months: number analyzed (Participants) | 118 | 101
  6 months | 9.3 (5.1) | 8.1 (5.2)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs PS-cCBT; Test type: Superiority; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected during the duration of the participants participation in the study, which in this case, was 6 months.
Arm/Group | Enhanced Usual Care | PS-cCBT
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/167
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/167
Other Adverse Events (participants affected / at risk) | 0/163 | 0/167

LIMITATIONS AND CAVEATS:
Follow-up assessment rates were lower than anticipated which may have reduced overall statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT02057042/Prot_SAP_000.pdf